CLINICAL TRIAL: NCT00841776
Title: Comparative Antimicrobial Efficacy of Two Topical Acne Therapies for the Treatment of Moderate to Moderately Severe Facial Acne Vulgaris
Brief Title: Comparative Antimicrobial Efficacy of Two Topical Acne Therapies for the Treatment of Facial Acne
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DTG0703
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Results first posted 2010-07-23 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Acne
Keywords: Acne Vulgaris; Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — clindamycin phosphate benzoyl peroxide combination

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duac gel (Active Comparator): Clindamycin and benzoyl peroxide gel
  Interventions: Drug: Duac
- Ziana gel (Active Comparator): Clindamycin and tretinoin gel
  Interventions: Drug: Ziana gel

INTERVENTIONS:
Drug: Duac — Clindamycon and benzoyl peroxide topical gel once a day for 12 weeks
  Arms: Duac gel
Drug: Ziana gel — Clindamycin and tretinoin gel once a day for 12 weeks.
  Arms: Ziana gel

SUMMARY:
The purpose of the study is to determine the development of microbial resistance when using one of two topical acne therapies for the treatment of facial acne vulgaris.

DETAILED DESCRIPTION:
To investigate the development of microbial resistance when using one of two topical acne therapies for the treatment of moderate to moderately severe facial acne vulgaris. Clinical efficacy and tolerability will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient at least 12 years of age. Female subjects of childbearing potential must have a negative urine pregnancy test result at baseline and practice a reliable method of contraception throughout the study.
* Mild to moderate facial acne vulgaris
* Able to understand the requirements of the study and sign informed consent/HIPAA authorization forms. Subjects under the legal age of consent in the state where the study is conducted must also have the written, informed consent of a parent or legal guardian.

Exclusion Criteria:

* Female subjects who are pregnant (positive urine pregnancy test), breast feeding or who are of childbearing potential and not practicing a reliable method of birth control
* Allergy or sensitivity to any component of the test medication
* Known hypersensitivity to to any component of the investigational formulations
* Known history of enteritis (regional enteritis, ulcerative colitis, pseudomembranous colitis, or antibiotic-associated colitis
* Beards or sideburns
* Skin disease/disorder that might interfere with the diagnosis or evaluation of acne vulgaris
* Evidence of recent alcohol or drug abuse
* Participation in an investigational drug study within 30 days of the baseline visit

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2007-08; Primary Completion 2008-11 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - Dermatology Specialists, PSC, Louisville, Kentucky
  - Skin We Care Dermatology, Mason, Ohio

REFERENCES:
- [Result] Jackson JM, Fu JJ, Almekinder JL. A randomized, investigator-blinded trial to assess the antimicrobial efficacy of a benzoyl peroxide 5%/ clindamycin phosphate 1% gel compared with a clindamycin phosphate 1.2%/tretinoin 0.025% gel in the topical treatment of acne vulgaris. J Drugs Dermatol. 2010 Feb;9(2):131-6. PMID 20214175

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Clinical research center
Groups:
- Duac: Clindamycin and benzoyl peroxide topical gel
- Ziana: Clindamycin and topical tretinoin gel
Period: Overall Study
Arm/Group | Duac | Ziana
Started | 27 | 27
Completed | 25 | 24
Not Completed | 2 | 3
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duac | Ziana | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.6 (6.9) | 16.2 (4.9) | 16.9 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 13 | 12 | 25
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 21 | 22 | 43
  Black | 4 | 4 | 8
  Hispanic | 0 | 1 | 1
  Other | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 27 | 27 | 54
Acne Lesion Counts [Mean (Standard Deviation); unit: Acne Lesion Counts] — P. acne Lesion Counts
  Acne Lesion Counts
    Inflammatory Lesion Counts | 24.74 (10.61) | 22.78 (7.07) | 23.76 (8.98)
    Noninflammatory Lesion Counts | 34.30 (20.38) | 35.11 (15.40) | 34.70 (17.90)
    Total Lesion Counts | 59.04 (23.68) | 57.89 (19.99) | 58.46 (21.72)
Clinidamycin-resistant propionibacterium acne (P.acne) counts [Mean (Standard Deviation); unit: Clinidamycin-resistant p. acne counts] — Clinidamycin-resistant Colony Forming Unit Propionibacterium acne counts
  Clinidamycin-resistant p. acne counts | 2.29 (1.34) | 2.02 (1.21) | 2.16 (1.27)
Erythromycin-resistant lesion count [Mean (Standard Deviation); unit: Erythromycin-resistant lesion count] — Erythromycin-resistant Colony forming Unit lesion count
  Erythromycin-resistant lesion count | 2.29 (1.37) | 1.92 (1.11) | 2.10 (1.25)
Propionibacterium acne counts [Mean (Standard Deviation); unit: P. acne counts] — Mean colony forming unit P. acne counts
  P. acne counts | 4.63 (1.12) | 4.74 (0.58) | 4.69 (0.88)

OUTCOME MEASURES:

1. Primary Outcome: Median Change in Total Propionibacterium Acne (P.Acne) Counts
Description: Median change in total colony forming units of propionibacterium acne (P.acne) will be counted.
Time Frame: Baseline, Weeks 2, 4, 8, 12, & 16
Measure: Median (Inter-Quartile Range); unit: P. acne counts
Arm/Group | Duac | Ziana
Number analyzed (Participants) | 27 | 27
P. acne counts
  Change from Baseline to Week 2 | -1.26 (1.44) [-2.42 to -0.4] | -0.08 (0.82) [-0.67 to 0.18]
  Change from Baseline to Week 4 | -1.58 (1.49) [-2.27 to -0.61] | -0.67 (1.18) [-1.31 to -0.04]
  Change from Baseline to Week 8 | -1.65 (1.50) [-2.43 to -0.68] | -0.32 (1.04) [-0.84 to 0.12]
  Change from Baseline to Week 12 | -1.82 (1.60) [-3.62 to -1.0] | -0.59 (0.99) [-1.07 to 0.07]
  Change from Baseline to Week 16 | -2.48 (1.77) [-3.08 to -0.82] | -0.57 (0.83) [-1.18 to -0.36]

2. Secondary Outcome: Median Change in Clindamycin Resistant P. Acne.
Description: Median change in total colony forming units of clindamycin resistant p. acne.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16
Population: ITT
Measure: Median (Inter-Quartile Range); unit: Clindamycin- resistant P. acne counts
Arm/Group | Duac | Ziana
Number analyzed (Participants) | 27 | 27
Clindamycin- resistant P. acne counts
  Change from Baseline to Week 2 | -0.30 [-1.74 to 0] | 0 [0 to 0.4]
  Change from Baseline to Week 4 | 0 [-1.43 to 0] | 0 [-0.51 to 0.12]
  Change from Baseline to Week 8 | -0.86 [-1.95 to 0] | 0 [-0.10 to 0.60]
  Change from Baseline to Week 12 | -0.83 [-1.53 to 0] | 0.39 [0 to 0.88]
  Change from Baseline to Week 16 | -0.30 [-1.84 to 0] | 0 [-0.03 to 0.25]

3. Secondary Outcome: Median Change in Erythromycin-resistant P. Acne Counts
Description: Total colony forming units of erythromycin-resistant p. acnes.
Time Frame: Baseline, Weeks 2, 4, 8, 12, and 16
Population: ITT
Measure: Median (Inter-Quartile Range); unit: Erythromycin-resistant P. acne counts
Arm/Group | Duac | Ziana
Number analyzed (Participants) | 27 | 27
Erythromycin-resistant P. acne counts
  Change from Baseline to Week 2 | -0.36 [-1.67 to 0] | 0 [0 to 0.56]
  Change from Baseline to Week 4 | -0.18 [-1.51 to 0] | 0 [0 to 0.68]
  Change from Baseline to Week 8 | -0.83 [-2.26 to 0] | 0 [0 to 0.40]
  Change from Baseline to Week 12 | -.91 [-1.68 to 0] | 0.15 [0 to 0.88]
  Change from Baseline to Week 16 | 0 [-1.81 to 0] | 0.04 [0 to 0.48]

4. Secondary Outcome: Median Change in Total Acne Lesions
Description: Median Change in Total Acne Lesions
Time Frame: Baseline, Weeks 2, 4, 8, 12, and 16
Population: ITT
Measure: Median (Inter-Quartile Range); unit: Total Acne Lesion Counts
Arm/Group | Duac | Ziana
Number analyzed (Participants) | 27 | 27
Total Acne Lesion Counts
  Change from Baseline to Week 2 | -14 [-22 to -4] | -13 [-23 to 2]
  Change from Baseline to Week 4 | -22 [-30 to -16] | -14 [-24 to -2]
  Change from Baseline to Week 8 | -27 [-38 to -9] | -19 [-36 to -5]
  Change from Baseline to Week 12 | -26.5 [-36 to -15] | -23.5 [-34 to -11]
  Change from Baseline to Week 16 | -33 [-35 to -22] | -30 [-41.5 to -17]

5. Secondary Outcome: Median Change in Inflammatory Acne Lesion Counts
Description: Median Change in Inflammatory Acne Lesion Counts
Time Frame: Baseline, Weeks 2, 4, 8, 12, and 16
Population: ITT
Measure: Median (Inter-Quartile Range); unit: Lesion Counts
Arm/Group | Duac | Ziana
Number analyzed (Participants) | 27 | 27
Lesion Counts
  Change from Baseline to Week 2 | -7 [-13 to -1] | -7 [-15 to -4]
  Change from Baseline to Week 4 | -12 [-18 to -3] | -7 [-15 to -1]
  Change from Baseline to Week 8 | -11 [-22 to -6] | -7 [-16 to -2]
  Change from Baseline to Week 12 | -12.5 [-19 to -7] | -10.5 [-17 to -5]
  Change from Baseline to Week 16 | -14 [-20 to -6] | -14 [-19 to -8]

6. Secondary Outcome: Median Change in Noninflammaotry Acne Counts
Description: Median Change in Noninflammaotry Acne Counts
Time Frame: Baseline, Weeks 2, 4, 8, 12, and 16
Measure: Median (Inter-Quartile Range); unit: Noninflammatory lesion counts
Arm/Group | Duac | Ziana
Number analyzed (Participants) | 27 | 27
Noninflammatory lesion counts
  Change from Baseline to Week 2 | -6 [-10 to 1] | -6 [-9 to 2]
  Change from Baseline to Week 4 | -10 [-23 to -3] | -8 [-18 to 1]
  Change from Baseline to Week 8 | -13 [-17 to -5] | -12 [-22 to 2]
  Change from Baseline to Week 12 | -9 [-25 to -4] | -13.5 [-18 to -2]
  Change from Baseline to Week 16 | -11 [-20 to -3] | -16.5 [-23 to -7.5]

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Duac | Ziana
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 5/27 | 5/27
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duac (N=27) | Ziana (N=27)
Attention Deficit Disorder (Nervous system disorders) | 1 (1) | 0 (0)
Sinus Infection (Infections and infestations) | 1 (1) | 1 (1)
Gonorrhea (Infections and infestations) | 1 (1) | 0 (0)
Head Cold (Infections and infestations) | 2 (3) | 1 (1)
Oral Thrush (Infections and infestations) | 1 (1) | 0 (0)
Oily skin on face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin surgery (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) — Surgery performed while on study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days